CLINICAL TRIAL: NCT04717219
Title: Myeloid Cell Reprogramming in Aortic Valve Stenosis
Brief Title: Myeloid Cells in Aortic Valve Stenosis
Acronym: MIRACLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Niels Riksen, Prof. dr., Radboud University Medical Center
Other Study IDs: NL72973.091.20
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis
Keywords: calcific aortic valve disease; valvular heart disease; inflammation; innate immune cells
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Heart Valve Diseases; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Severe CAVD with atherosclerosis: Participants with severe CAVD and significant atherosclerosis
  Interventions: Other: Blood drawing
- Severe CAVS without atherosclerosis: Participants with severe CAVD without significant atherosclerosis
  Interventions: Other: Blood drawing
- Moderate CAVD with atherosclerosis: Participants with mild or moderate CAVD and significant atherosclerosis
  Interventions: Other: Blood drawing
- Moderate CAVD without atherosclerosis: Participants with mild or moderate CAVD without significant atherosclerosis
  Interventions: Other: Blood drawing
- Healthy controls: Healthy controls without CAVD and without a history of atherosclerotic cardiovascular events, current typical complaints of angina pectoris or intermittent claudication and overt heart failure (NYHA class III/IV).
  Interventions: Other: Blood drawing
- Controls with bicuspid aortic valve stenosis: Controls with bicuspid aortic valve stenosis, without a history of atherosclerotic cardiovascular events, current typical complaints of angina pectoris or intermittent claudication.
  Interventions: Other: Blood drawing

INTERVENTIONS:
Other: Blood drawing — Blood will be drawn after inclusion of the participants.

SUMMARY:
Investigators plan to characterize systemic inflammation and circulating immune cells in participants with moderate and severe calcific aortic valve disease and matched healthy controls.

DETAILED DESCRIPTION:
Calcific aortic valve disease (CAVD) is the most common type of valvular heart disease in the Western world. Due to the aging of the population, the impact of this disorder is expected to further increase in the next decades. The underlying pathophysiology remains incompletely defined and there are currently no effective medical treatments capable of altering its course, identifying a major unmet need in this growing population of patients.

Based on the similarities between CAVD and atherosclerosis in pathophysiology and shared risk factors, it is now hypothesized that activation of the innate immune system contributes to the development of CAVD. Therefore, the investigators will perform an observational study to assess the role of activation of the innate immune system in CAVD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mild, moderate or severe degenerative aortic valve stenosis as defined by transthoracic echocardiography according to the 2017 ESC/EACTS guidelines for the management of valvular heart disease.

Exclusion Criteria:

* Active auto-inflammatory or auto-immune diseases
* Anti-inflammatory drugs
* Vaccination less than one month before inclusion
* Bone marrow transplantation
* Active malignancy, except for local basal cell carcinoma or local squamous cell skin carcinoma, that can be treated curatively by excision.
* History of endocarditis of the aortic valve
* History of radiation therapy aimed at the chest
* Acute ischemic cardiac event less than three months before inclusion
* Systemic inflammation less than one month before inclusion with fever and/or for which antibiotics have been prescribed, with the exception for the use of nitrofurantoin for a urinary tract infection without fever

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present themselves or are already known at the department of cardiology or cardiothoracic surgery with the diagnosis of moderate or severe aortic valve stenosis as defined by transthoracic echocardiography according to the 2017 ESC/EACTS guidelines for the management of valvular heart disease.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammatory phenotype of circulating immune cells. | 2 years
  The inflammatory phenotype of circulating immune cells will be measured by determining the cytokine production capacity after stimulation with relevant stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Niels P. Riksen, prof. dr., Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Rijnstate, Arnhem
  - Radboud university medical center, Nijmegen
  - Canisius Wilhelmina Ziekenhuis, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided